CLINICAL TRIAL: NCT02396303
Title: Carbetocin Versus Oxytocin in Caesarean Section for the Control of Postpartum Haemorrhage
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Mousumi Paul, FCPS Course Student, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 67365
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Postpartum Haemorrhage
Keywords: General: To compare Carbetocin and Oxytocin for the control of PPH.
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient receiving carbetocin (Experimental): Experimental group subjects will receive intravenous Carbetocin during third stage of labour.
  Interventions: Drug: Carbetocin
- Patient receiving oxytocin (Active Comparator): Comparator group subjects will receive intramascular Oxytocin during third stage of labour.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin

SUMMARY:
Post-partum haemorrhage is one of the life threatening emergencies. It accounts for nearly one-quarter of all maternal death worldwide. Atonic uterus contributes about 80% among the causes. Uterotonic drugs are administered following the delivery of baby both in vaginal and caesarean delivery for prevention of PPH. However postpartum haemorrhage cannot always be prevented. But, the incidence and especially its magnitude can be reduced by assessing the risk factors and following the guidelines. The intelligent anticipation, skilled supervision, prompt detection and effective institution of therapy can prevent a normal case from undergoing disastrous consequences. This study will be carried out at Bangabandhu Sheikh Mujib Medical University (BSMMU) within six months after approval. This is a Randomized Control Trial which will compare efficacy of Carbetocin and Oxytocin for the control of PPH. Structured Questionnaire, Data Sheet, hospital indoor documents i.e. Patient chart, operation notes, surgeons visual estimation of blood loss etc will be used as study tool. Ethical clearance will be obtained from Institutional Review Board of BSMMU. Written informed consent will be obtained from the patient or from her legal guardian. Patient confidentiality will be strictly maintained. No name, address or contact details of the patient will be divulged.

ELIGIBILITY:
Inclusion Criteria:

* Patient with risk factors for primary post-partum haemorrhage such as: multiple pregnancy, one or more previous caesarean section, presence of uterine fibroids, previous myomectomy, presence of placenta previa, past history of PPH, fetal macrosomia and fetal malformations associated with polyhydramnios

Exclusion Criteria:

* Presence of hypertension, eclampsia, cardiac, renal or liver diseases, epilepsy, general anaesthesia, as well as women with history of hypersensitivity to Carbetocin according to the Br National Formulary. Patients unwilling to give consent for this study are also excluded

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-10 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Estimated blood loss after cesarean section | 24 hours of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- BSMMU, Dhaka, Bangladesh